CLINICAL TRIAL: NCT01625611
Title: Kappa-PET Imaging and Naltrexone in Alcohol Drinking Behaviors
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Yale University (Other)
Collaborators: National Institute on Alcohol Abuse and Alcoholism (NIAAA) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 1011007710; R01AA021818-01A1 (NIH); U54AA027989 (NIH)
Record Dates: First submitted 2012-06-19; First posted 2012-06-21 (Estimated); Results first posted 2022-08-10 (Actual); Last update posted 2022-08-10 (Actual); Status verified 2022-08

CONDITIONS: Alcohol Drinking
Keywords: Alcohol; Drinking; Drinkers; Alcohol Drinking; Naltrexone; Alcohol Dependence; Alcohol Abuse; Alcohol-Related Disorders; Ethanol; Alcoholism
MeSH Terms: conditions — Alcohol Drinking; Alcoholism; Alcohol-Related Disorders | interventions — Naltrexone

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Naltrexone (Experimental)
  Interventions: Drug: Naltrexone

INTERVENTIONS:
Drug: Naltrexone — Naltrexone 100 mg titrated over one week
  Other Names: Revia

SUMMARY:
The primary purpose of the study is to increase our knowledge of receptor function in the brains of people who are heavy drinkers and taking naltrexone (NTX), a medication that has been approved for the treatment of alcohol dependence. Receptors are special molecules in the brain to which other molecules (neurotransmitters) attach during the normal every-day workings of the brain. Drugs can bind to those receptor molecules as well. Recent evidence suggests that kappa opioid receptors (KOR's) may play an important role in alcohol drinking behavior. This study will try to determine if naltrexone's ability to attach to these receptors is related to its effectiveness. We will use PET (positron emission tomography) for this study. PET is a type of imaging device found in nuclear medicine. It is used for tracking the presence of injected radioactive materials in the body.

ELIGIBILITY:
Inclusion Criteria:

* Ages 21-50
* Able to read English at 6th grade level or higher and to complete study evaluations
* Regular alcohol drinker

Exclusion Criteria:

* Individuals who are seeking alcohol treatment
* Medical conditions that would contraindicate the use of study medication
* Regular use of other substances

Ages: 21 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 59 (Actual)
Dates: Start 2011-02; Primary Completion 2021-06-30 (Actual); Study Completion 2021-06-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Suchitra Krishnan-Sarin, Ph.D., Principal Investigator — Yale University
Locations (1):
- Sac, Cmhc, New Haven, Connecticut, United States

REFERENCES:
- [Derived] de Laat B, Goldberg A, Shi J, Tetrault JM, Nabulsi N, Zheng MQ, Najafzadeh S, Gao H, Kapinos M, Ropchan J, O'Malley SS, Huang Y, Morris ED, Krishnan-Sarin S. The Kappa Opioid Receptor Is Associated With Naltrexone-Induced Reduction of Drinking and Craving. Biol Psychiatry. 2019 Dec 1;86(11):864-871. doi: 10.1016/j.biopsych.2019.05.021. Epub 2019 Jun 8. PMID 31399255

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were recruited from the community through various methods such as flyers and online.
Pre-assignment Details: All enrolled participants were assigned to a study arm.
Groups:
- Healthy Controls: No treatment, baseline measurements only.
Period: Overall Study
Arm/Group | Naltrexone | Healthy Controls
Started | 55 | 4
PET Scan 1 | 49 | 4
Lab 2 | 48 | 0
PET Scan 2 | 47 | 0
Completed | 47 | 4
Not Completed | 8 | 0
Not completed — No adlib drinks Lab 1 | 3 | 0
Not completed — Technical issues with PET | 1 | 0
Not completed — Unable to complete study procedures | 1 | 0
Not completed — Withdrawal by Subject | 3 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Naltrexone | Healthy Controls | Total
Number analyzed (Participants) | 47 | 4 | 51
Age, Continuous [Mean (Standard Deviation); unit: years] | 32 (3.9) | 35.6 (11.4) | 33.8 (7.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 16 | 3 | 19
  Male | 31 | 1 | 32
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 8 | 0 | 8
  Not Hispanic or Latino | 39 | 4 | 43
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 22 | 0 | 22
  White | 24 | 4 | 28
  More than one race | 1 | 0 | 1
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 47 | 4 | 51

OUTCOME MEASURES:

1. Primary Outcome: Occupancy of KOR by NTX and Drinking
Description: To determine the degree to which occupancy of KORs by a 100 mg/day dose of NTX mediates (influences the strength of) responsivity to NTX treatment in all heavy drinkers.
Time Frame: 6-8 days after treatment with naltrexone
Measure: Mean (Standard Error); unit: % Occupancy
Arm/Group | Naltrexone
Number analyzed (Participants) | 44
% Occupancy | 92 (1)

2. Primary Outcome: Relationship Between NTX Responsivity and Occupancy of KOR
Description: To determine whether the relationship between NTX responsivity and occupancy of KOR is different in family history positive vs. family history negative heavy drinkers. Evaluations were done with a logistic regression which included years of drinking (a covariate), family history status, and occupancy of KOR. The logistic model calculated a probability of response, defined as a 50% or greater reduction in drinking after naltrexone, for every participant. Reported outcome is the area under the ROC produced by the model. The closer the value is to 100 percent probability, the better the model is at correctly classifying the observations.
Time Frame: 6-8 days after treatment with naltrexone
Measure: Number; unit: percent probability
Arm/Group | Naltrexone
Number analyzed (Participants) | 44
percent probability | 84

3. Secondary Outcome: Baseline KOR Differences
Description: To determine if baseline levels of KOR differ between family history positive (FHP) and family history negative (FHN) heavy drinkers and to determine if baseline KOR level is related to either baseline drinking or responsivity to NTX.
Time Frame: at baseline prior to treatment with naltrexone
Measure: Mean (Standard Error); unit: % Occupancy
Groups:
- Naltrexone - FH Positive; Naltrexone - FH Negative: Naltrexone: Naltrexone 100 mg titrated over one week
Arm/Group | Naltrexone - FH Positive | Naltrexone - FH Negative
Number analyzed (Participants) | 29 | 18
% Occupancy | 91.2 (1.7) | 94.2 (1.9)

ADVERSE EVENTS:
Time Frame: Approximately 3 weeks
Arm/Group | Naltrexone | Healthy Controls
All-Cause Mortality (participants affected / at risk) | 0/55 | 0/4
Serious Adverse Events (participants affected / at risk) | 0/55 | 0/4
Other Adverse Events (participants affected / at risk) | 37/55 | 0/4
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Naltrexone (N=55) | Healthy Controls (N=4)
Nausea (Gastrointestinal disorders) | 19 (22) | 0 (0)
Vomiting (Gastrointestinal disorders) | 6 (7) | 0 (0)
Diarrhea (Gastrointestinal disorders) | 6 (7) | 0 (0)
Abdominal discomfort (Gastrointestinal disorders) | 3 (3) | 0 (0)
Headache (Nervous system disorders) | 9 (10) | 0 (0)
Fatigue (General disorders) | 4 (4) | 0 (0)
Anxiety (Psychiatric disorders) | 3 (3) | 0 (0)
Insomnia (General disorders) | 1 (1) | 0 (0)
Drowsiness (General disorders) | 2 (3) | 0 (0)
Depression (Psychiatric disorders) | 1 (1) | 0 (0)
Cloudy (General disorders) | 1 (1) | 0 (0)
Cold sweat (General disorders) | 1 (1) | 0 (0)
Congestion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Hypothermia (General disorders) | 1 (1) | 0 (0)
Constipation (Gastrointestinal disorders) | 2 (2) | 0 (0)
Decreased desired to drink (General disorders) | 1 (1) | 0 (0)
Decreased sex drive (Reproductive system and breast disorders) | 3 (3) | 0 (0)
Dry mouth (Gastrointestinal disorders) | 1 (1) | 0 (0)
Feeling high (General disorders) | 3 (3) | 0 (0)
Feeling good (General disorders) | 1 (2) | 0 (0)
Frequent urination (Renal and urinary disorders) | 3 (3) | 0 (0)
Irritability (Psychiatric disorders) | 1 (2) | 0 (0)
Muscle tightness (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Peeling hands (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Tremor (Nervous system disorders) | 2 (2) | 0 (0)
Stomach ache (Gastrointestinal disorders) | 1 (1) | 0 (0)
Tightness in chest (General disorders) | 1 (1) | 0 (0)
Tired (General disorders) | 3 (3) | 0 (0)
Upset stomach (Gastrointestinal disorders) | 1 (2) | 0 (0)
Apetite change (Gastrointestinal disorders) | 5 (5) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (3):
  • Study Protocol and Statistical Analysis Plan (2019-05-06): https://cdn.clinicaltrials.gov/large-docs/11/NCT01625611/Prot_SAP_000.pdf
  • Informed Consent Form: Naltrexone group (2018-01-10): https://cdn.clinicaltrials.gov/large-docs/11/NCT01625611/ICF_001.pdf
  • Informed Consent Form: Healthy control group (2018-01-10): https://cdn.clinicaltrials.gov/large-docs/11/NCT01625611/ICF_002.pdf